CLINICAL TRIAL: NCT03011710
Title: Epidemiology and Acute Oral Effects of Electronic Cigarette
Brief Title: Epidemiology and Acute Oral Effects Electronic Cigarette
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: epidacute-ecig-2015
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2022-07

CONDITIONS: Nicotine Dependence, Cigarettes
Keywords: e-cigarette; blood flow; oral effects; oral pH
MeSH Terms: conditions — Tobacco Use Disorder; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- E-cigarette with nicotine (Experimental): Nicotine level: 6 mg/ml
  Interventions: Device: ProVari v2.5 (E-cigarette)
- E-cigarette without nicotine (Experimental): Nicotine level: 0 mg/ml
  Interventions: Device: ProVari v2.5 (E-cigarette)
- Conventional cigarette (Experimental): Nicotine content: 0,5mg
  Interventions: Device: Marlboro Gold (Conventional cigarette)
- Cigarette tip (Placebo Comparator): Placebo device
  Interventions: Device: Cigarette tip

INTERVENTIONS:
Device: ProVari v2.5 (E-cigarette) — An electronic cigarette or e-cigarette is a handheld electronic device that vaporizes a flavored liquid. The user inhales the vapor. The fluid in the e-cigarette, called e-liquid, is usually made of nicotine, propylene glycol, glycerine, and flavorings.
  Other Names: ProVari v2.5
  Arms: E-cigarette with nicotine; E-cigarette without nicotine
Device: Marlboro Gold (Conventional cigarette) — Conventional cigarette
  Other Names: Marlboro Gold 0,6mg
  Arms: Conventional cigarette
Device: Cigarette tip — Placebo device
  Arms: Cigarette tip

SUMMARY:
Electronic cigarettes are battery-powered vaporizers which have a similar feel to tobacco smoking. They do not produce cigarette smoke but rather an aerosol, which is frequently referred to as vapor. E-cigarettes are marketed as less harmful alternatives to smoking. Use and awareness of these devices has grown exponentially in recent years, with millions of people currently using them.

The benefits and risks of electronic cigarette use are uncertain. There is no research on the acute oral effects of electronic cigarette in the scientific literature and no hungarian epidemiological survey has been performed in this topic.

Regulation of electronic cigarettes varies across countries in the European Union, ranging from no regulation to banning them entirely.

The investigators research could help to integrate the regulation of this device in Hungary and in the EU as well.

The measurement of acute oral effects of e-cigarette and a hungarian epidemiological survey would be novel in this topic.

DETAILED DESCRIPTION:
The epidemiological survey is performed with online questionnaires, which are published on e-cigarette-selling websites and on other forums dealing with this topic.

The main outcome of interest was whether or not e-cigarette use helped people to quit smoking or reduce the number of conventional cigarettes. Participants were also asked about the reason for starting e-cigarette use. Nationality, habitation, citizenship status were included as demographic predictors in analyses.

Measurements of acute oral effects before and after using electronic cigarette with nicotine, without nicotine, conventional cigarette and placebo device:

* measurement of exhaled CO changes by Smokerlyzer piCO
* measurement of saliva MMP-8 by PerioSafe Home
* measurement of saliva pH, buffering capacity, and flow rate changes by Saliva Check Buffer Kit (GC)
* measurement of oral mucosal blood flow changes by Perilam PSI System High Resolution (LASCA method)

ELIGIBILITY:
Inclusion Criteria:

* age: 19-49 years
* signed consent form
* smoking regularly e-cigarette and/or conventional cigarette for > half year

Exclusion Criteria:

* not pregnant and not planning pregnancy in the next 6 month
* BMI index < 30
* no severe parodontal disease
* no acute illness in the last 2 weeks
* no chronic disease (eg.: diabetes)
* no diet which can influence the oral pH

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-09; Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood flow after vaping/smoking | baseline, immediately after smoking/vaping, and 15 minutes after smoking/vaping
  The blood flow changes are measured by Laser Speckle Contrast Analyzer (LASCA) before (baseline) and after vaping/smoking.

IPD SHARING:
Plan to Share IPD: No